CLINICAL TRIAL: NCT07151105
Title: Anti-inflammatory Activities of Vitamin C Supplementation on the Gut Barrier Function in Adults With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY20251283
Record Dates: First submitted 2025-08-27; First posted 2025-09-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Adequate Vitamin C Status; Inadequate Vitamin C Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inadequate Vitamin C Status (Placebo Comparator): Placebo + Low Vitamin C Diet
  Interventions: Dietary Supplement: Placebo + Low Vitamin C Diet
- Adequate Vitamin C Status (Experimental): Vitamin C Supplement + Low Vitamin C Diet
  Interventions: Dietary Supplement: Vitamin C Supplement + Low Vitamin C Diet

INTERVENTIONS:
Dietary Supplement: Vitamin C Supplement + Low Vitamin C Diet — Participants will receive a vitamin C supplement (1000 mg/d) while following a low vitamin C diet to achieve adequate vitamin C status in a blinded manner. This will be compared to participants receiving a placebo while following a low vitamin C diet that is expected to maintain inadequate vitamin C status.
  Arms: Adequate Vitamin C Status
Dietary Supplement: Placebo + Low Vitamin C Diet — Participants will receive a placebo while following a low vitamin C diet to achieve inadequate vitamin C status in a blinded manner. This will be compared to participants receiving a vitamin C supplement while following a low vitamin C diet that is expected to maintain adequate vitamin C status.
  Arms: Inadequate Vitamin C Status

SUMMARY:
This study is testing whether taking vitamin C every day can help improve gut health and reduce inflammation in adults with obesity. Poor gut health-sometimes called "leaky gut"-can allow harmful substances from bacteria to enter the bloodstream, which may lead to inflammation and increase the risk of heart disease and liver problems.

Participants will complete two study periods, each lasting two weeks, with a two-week break in between. In one period, they will take vitamin C; in the other, a placebo. During each period, researchers will collect blood, urine, and stool samples, ask participants to track their diet and activity, and perform a test to measure gut permeability.

There are minimal risks, such as discomfort from blood draws or temporary stomach upset from a sugar drink. While participants may not directly benefit, their involvement will help researchers learn whether vitamin C is a safe and effective way to improve gut health in people with obesity.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the impact of vitamin C supplementation on gut barrier function and systemic inflammation in adults with obesity. The research builds on preclinical findings that suggest vitamin C plays a critical role in maintaining gut integrity and reducing inflammation. Approximately 40% of Americans have suboptimal vitamin C status, with even higher prevalence among individuals with obesity.

The primary hypothesis is that improving vitamin C status through dietary supplementation will reduce intestinal permeability and metabolic endotoxemia. A secondary hypothesis is that vitamin C will also reduce biomarkers of intestinal inflammation and promote favorable changes in gut microbiota composition, including increased production of short-chain fatty acids (SCFAs), which are essential for intestinal health.

This randomized, double-blind, placebo-controlled crossover trial will enroll 34 obese adults (BMI 30-40 kg/m², aged 18-50 years). Participants will complete two 2-week intervention periods separated by a 2-week washout. In one period, they will receive vitamin C (500 mg capsules taken twice daily); in the other, a placebo. During both periods, participants will follow a low-vitamin C diet to minimize variability in circulating vitamin C levels.

Assessments will occur on Days 0, 7, and 14 of each intervention period and include: Anthropometric measurements; Resting blood pressure; Fasting blood samples; and 3-day food records. On Day 14 of each period, participants will: Provide a stool sample and Complete a gut permeability test using a non-digestible sugar probe solution followed by a 24-hour urine collection. After the first intervention period, participants will undergo a 2-week washout before repeating the procedures with the alternate supplement.

Primary Outcome: Intestinal permeability

Secondary Outcomes: Biomarkers of endotoxemia; Gut microbiota composition; Intestinal and circulating inflammation biomarkers; Plasma vitamin C concentrations; Fecal short-chain fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Men and women between 18-50 years of age
* BMI 30-40 kg/m²
* Resting blood pressure <140/90 mm Hg
* No use of multivitamin/vitamin C supplement within past 1-month
* Non-vegetarian/non-vegan
* Willingness to follow a diet low in fruits and vegetables for two, 2-week periods

Exclusion Criteria:

* Current smoker or vaper, including tobacco, cannabis, or nicotine products
* Alcohol consumption >2 drinks/day
* Use of antibiotics within past 1-month
* Use of probiotic supplements within past 1-month
* Use of anti-inflammatory drugs within past 1-month
* Individuals with unmanaged or poorly controlled diabetes, dyslipidemia, hypertension
* Known history of bleeding disorders, hemochromatosis, or kidney stones
* For Women: Pregnancy, lactation, or change in birth control within the past 3-months
* Use of certain medications that may interact with vitamin C, including blood thinners, some antiviral drugs (e.g., indinavir), and certain antipsychotic medications (e.g., fluphenazine).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Small Intestinal Permeability | Between-treatment arm comparison on day 14 following 2-week intervention.
  Urinary excretion ratio of lactulose/mannitol following oral ingestion of these sugar probes.

SECONDARY OUTCOMES:
Large Intestinal Permeability | Between-treatment arm comparison on day 14 following 2-week intervention.
  Urinary excretion ratio of sucralose/erythritol following oral ingestion of these sugar probes.
Plasma Vitamin C | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Vitamin C
Plasma Vitamin C | Within-treatment arm comparison from day 0 to day 14 following 2-week intervention.
  Biochemical measures of Vitamin C
Fecal Calprotectin | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Calprotectin
Fecal Myeloperoxidase | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Myeloperoxidase
Fecal Butyrate | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Butyrate
Fecal Proprionate | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Proprionate
Fecal Acetate | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Acetate
Serum Endotoxin Concentration | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measure of circulating endotoxin concentration at fasting
Plasma Lipopolysaccharide Binding Protein/Soluble Cluster of Differentiation-14 | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Lipopolysaccharide Binding Protein/Soluble Cluster of Differentiation-14 at fasting, reported as a ratio of protein concentrations
Plasma C-Reactive Protein | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of C-Reactive Protein
Plasma Myeloperoxidase | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Myeloperoxidase
Plasma Tumor Necrosis Factor-α | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Tumor Necrosis Factor-α
Plasma Trimethylamine N-oxide | Between-treatment arm comparison on day 14 following 2-week intervention.
  Biochemical measures of Trimethylamine N-oxide

OTHER OUTCOMES:
alpha-Diversity (Chao1) | Between-treatment arm comparison on day 14 following 2-week intervention
  Gut microbiota alpha-diversity will be determined from 16S rRNA sequencing
alpha-Diversity (Shannon Index) | Between-treatment arm comparison on day 14 following 2-week intervention
  Gut microbiota alpha-diversity will be determined from 16S rRNA sequencing
beta-Diversity (Bray-Curtis Dissimilarity) | Between-treatment arm comparison on day 14 following 2-week intervention
  Gut microbiota beta-diversity will be determined from 16S rRNA sequencing
beta-Diversity (UniFrac) | Between-treatment arm comparison on day 14 following 2-week intervention
  Gut microbiota beta-diversity will be determined from 16S rRNA sequencing
Toll-like Receptor-4 mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood
TNF-alpha mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood
Monocyte Chemoattract Protein-1 mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood
Interleukin-6 mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood
Interleukin-8 mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood
Myeloid differentiation primary response 88 mRNA expression | Between-treatment arm comparison on day 14 following 2-week intervention.
  qPCR measure of gene expression from Peripheral Blood Mononuclear Cells isolated from whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Although no formal plan for sharing is established, data will be shared upon reasonable request and when in accordance with regulatory compliance considerations.

REFERENCES:
- [Background] Traber MG, Buettner GR, Bruno RS. The relationship between vitamin C status, the gut-liver axis, and metabolic syndrome. Redox Biol. 2019 Feb;21:101091. doi: 10.1016/j.redox.2018.101091. Epub 2018 Dec 26. PMID 30640128